CLINICAL TRIAL: NCT05147532
Title: Remyelination in Multiple Sclerosis: a PET-MR Longitudinal Study Investigating Individual Profiles of Myelin Repair and the Contribution of Neuroinflammation
Acronym: SMARTinMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP200056; 2021-002334-16 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2021-12-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Inflammatory Disease
Keywords: Multiple sclerosis; Remyelination; Combination of magnetic resonance imaging (MRI) and positron emission tomography (PET)
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-MRI with [18F]-Florbetaben and PET-MRI with [18F]-DPA-714 (Other): PET-MRI with [18F]-Florbetaben and PET-MRI with [18F]-DPA-714
  Interventions: Procedure: PET-MRI with [18F]-Florbetaben and PET-MRI with [18F]-DPA-714

INTERVENTIONS:
Procedure: PET-MRI with [18F]-Florbetaben and PET-MRI with [18F]-DPA-714 — PET-MRI: 2 at baseline visits (V0 and V1) and 1 at M6

SUMMARY:
Multiple Sclerosis (MS) is an inflammatory disease where the immune cells invade the central nervous system and destroy an essential element of nerve conduction: the myelin. An interesting feature observed in some patients is a regenerative process, called remyelination, which leads to the production of new myelin. However, the extent of remyelination is very heterogeneous among patients, only a minority of patients show a really efficient repair process along the disease course. In this project, our aim is to explore in vivo the biological mechanisms leading to a successful remyelination in some patients and to a failure in remyelination in others. With this purpose in mind we propose to develop a translational research platform where patients with multiple sclerosis will be investigated in vivo for their potential of remyelination through a follow-up with recently developed imaging technologies using a synergistic combination of magnetic resonance imaging (MRI) and positron emission tomography (PET) to visualize and quantify myelin and neuroinflammation. In parallel blood immune cells from patients will be sampled and profiled to investigate how they could influence remyelination. This part will consist in i) grafting patients' lymphocytes in experimental rodent models of demyelination to characterize how they could promote or inhibit remyelination; ii) performing a functional and multi-omics analysis of peripheral macrophages and analyse relationships with remyelination profiles; iii) profiling T lymphocytes at the single cell level to associate specific subpopulation of the T cells with the remyelination potential assessed in patients with MRI/PET images and in grafted animals.

ELIGIBILITY:
Inclusion Criteria:

RRMS patients:

1. Age between 18 and 55 years old
2. RRMS according to the 2017 Mc Donald criteria
3. Less than 5 years of disease duration
4. At least 9 supra-tentorial white matter lesions on T2/FLAIR MRI
5. Last treatment with methylprednisolone should have been performed at least 1 month before PET examinations
6. Interferon-beta, glatiramere acetate and oral first line therapy will such as dimethylfumarate or teriflunomide will be admitted
7. Affiliation to a social security scheme or beneficiary of such a scheme (Except "Aide Médicale d'Etat")

Progressive MS patients:

1. Age between 18 and 55 years old
2. Progressive MS (primary or secondary progressive MS) according to the 2017 Mc Donald criteria
3. Less than 10 years of disease duration in the progressive phase
4. At least 9 supra-tentorial white matter lesions on T2/FLAIR MRI
5. Interferon-beta, glatiramere acetate and oral first line therapy will such as dimethylfumarate or teriflunomide will be admitted
6. Affiliation to a social security scheme or beneficiary of such a scheme (except "Aide Médicale d'Etat")

Healthy volunteers:

1. Age between 18 and 55 years old
2. Without any evolutive pathology
3. Able to understand the study objectives and procedures
4. Affiliation to a social security scheme or beneficiary of such a scheme (except "Aide Médicale d'Etat")

Exclusion Criteria:

For all participants:

1. Any reasons, which does not allow to perform MRI, including claustrophobia, the implant of a pace maker or the presence of an intra-ocular foreign body (a contra-indication questionnaire will be filled in beforehand)
2. PET for clinical research already done within the last 12 months
3. Low Affinity Binding profile (TSPO polymorphism analyzed at screening visit)
4. Pregnancy, breast-feeding, lack of efficient contraception
5. Current symptoms of severe or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary or cardiac disease, or any other chronic neurological diseases
6. Unwillingness to be informed in case of abnormal MRI (with a significant medical anomaly)
7. Know hypersensitivity to Myelin PET : [18F]-Florbetaben
8. Patient under legal protection

Additional exclusion criteria for patients:

1. Treatment with cyclophosphamide, mitoxantrone, fingolimod, cladribine, alemtuzumab, anti CD20 antibodies or natalizumab will not be admitted. These treatments may be administered after the Baseline visit.
2. Known allergy to gadoteric acid
3. Allergies (seafood, pollinosis, urticarial) having required a medical intervention
4. Severe renal insufficiency (creatinine clearance < 60mL/min).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of lesional demyelinated voxels at baseline that are classified as remyelinating at month 6 of multiple sclerosis patients during the relapsing and the progressive phases of the disease | Month 6
  the percentage of lesional voxels classified as demyelinated on baseline [18F]-Florbetaben PET, that subsequently become normally myelinated on the [18F]-Florbetaben PET performed at 6 months, which attest remyelination

SECONDARY OUTCOMES:
the percentage of voxels classified as significantly activated compared to control white matter, and the number/proportion of MS lesions classified as activated based on [18F]-DPA-714 PET | At baseline
  To define the individual inflammatory profiles from [18F]-DPA-714 PET (regional individual maps of [18F]-DPA-714 binding) of MS patients during the relapsing and the progressive phases of the disease
Proportion of each lymphocyte cluster identified from the single cell sequencing of T lymphocytes over the total T lymphocyte population for each patient | Baseline
Remyelination level in rodents demyelinated by lysolecithin and grafted with single patient's lymphocytes quantified at week 3 post-graft | Baseline
Proportion of lesions that persist as chronic active at month 3 post graft over the total number of lesions induced in the rodent demyelinating models by grafting patients' lymphocytes | Baseline, at 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Neurosciences - Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodini B, Tonietto M, Airas L, Stankoff B. Positron emission tomography in multiple sclerosis - straight to the target. Nat Rev Neurol. 2021 Nov;17(11):663-675. doi: 10.1038/s41582-021-00537-1. Epub 2021 Sep 20. PMID 34545219
- [Background] Poirion E, Tonietto M, Lejeune FX, Ricigliano VAG, Boudot de la Motte M, Benoit C, Bera G, Kuhnast B, Bottlaender M, Bodini B, Stankoff B. Structural and Clinical Correlates of a Periventricular Gradient of Neuroinflammation in Multiple Sclerosis. Neurology. 2021 Apr 6;96(14):e1865-e1875. doi: 10.1212/WNL.0000000000011700. Epub 2021 Mar 18. PMID 33737372
- [Background] Auvity S, Tonietto M, Caille F, Bodini B, Bottlaender M, Tournier N, Kuhnast B, Stankoff B. Repurposing radiotracers for myelin imaging: a study comparing 18F-florbetaben, 18F-florbetapir, 18F-flutemetamol,11C-MeDAS, and 11C-PiB. Eur J Nucl Med Mol Imaging. 2020 Feb;47(2):490-501. doi: 10.1007/s00259-019-04516-z. Epub 2019 Nov 4. PMID 31686177
- [Background] Stankoff B, Poirion E, Tonietto M, Bodini B. Exploring the heterogeneity of MS lesions using positron emission tomography: a reappraisal of their contribution to disability. Brain Pathol. 2018 Sep;28(5):723-734. doi: 10.1111/bpa.12641. PMID 30020560
- [Background] Bodini B, Veronese M, Garcia-Lorenzo D, Battaglini M, Poirion E, Chardain A, Freeman L, Louapre C, Tchikviladze M, Papeix C, Dolle F, Zalc B, Lubetzki C, Bottlaender M, Turkheimer F, Stankoff B. Dynamic Imaging of Individual Remyelination Profiles in Multiple Sclerosis. Ann Neurol. 2016 May;79(5):726-738. doi: 10.1002/ana.24620. PMID 26891452
- [Background] Stankoff B, Freeman L, Aigrot MS, Chardain A, Dolle F, Williams A, Galanaud D, Armand L, Lehericy S, Lubetzki C, Zalc B, Bottlaender M. Imaging central nervous system myelin by positron emission tomography in multiple sclerosis using [methyl-(1)(1)C]-2-(4'-methylaminophenyl)- 6-hydroxybenzothiazole. Ann Neurol. 2011 Apr;69(4):673-80. doi: 10.1002/ana.22320. Epub 2011 Feb 18. PMID 21337603